CLINICAL TRIAL: NCT00869232
Title: UARK 2008-02, A Phase II Trial for High-risk Myeloma Evaluation Accelerating and Sustaining Complete Remission (AS-CR) by Applying Non-host-exhausting and Timely Dose-reduced MEL-80-VRD-PACE Tandem Transplants
Brief Title: UARK 2008-02 A Trial for High-risk Myeloma Evaluating Accelerating and Sustaining Complete Remission
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 106952
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Thalidomide; Dexamethasone; Calcium Dobesilate; Cisplatin; Doxorubicin; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MEL--VTD-PACE (Experimental): Melphalan, Velcade, Thalidomide, Dexamethasone, Cisplatin, Adriamycin, Cyclophosphamide and Etoposide
  Interventions: Drug: Velcade; Drug: Melphalan; Drug: Thalidomide; Drug: Dexamethasone; Drug: Cisplatin; Drug: Adriamycin; Drug: Cyclophosphamide; Drug: Etoposide

INTERVENTIONS:
Drug: Velcade — 1.0mg/m2 days 1, 5, 8, & 11
  Other Names: PS-341
Drug: Melphalan — 10 mg/m2 day 3
  Other Names: Alkeran
Drug: Thalidomide — 200 mg days 5-8
  Other Names: Thalomid
Drug: Dexamethasone — 40 mg day 5-8
  Other Names: Decadron
Drug: Cisplatin — 10 mg/m2 day 5-8
  Other Names: Platinol
Drug: Adriamycin — 10 mg/m2 day 5-8
  Other Names: Doxorubicin
Drug: Cyclophosphamide — 400 mg/m2 day 5-8
  Other Names: Cytoxan
Drug: Etoposide — 40 mg/m2 day 5-8
  Other Names: Vp-16, Vepesid

SUMMARY:
There have been four previous Total Therapy (TT1 through IIIB) studies for multiple myeloma at the MIRT from 1989 to present. Results have shown that participants treated on these studies had better outcomes (meaning they have lived longer and had better responses to treatment) when compared to individuals treated with standard chemotherapy.

Past studies conducted at the MIRT and at other institutions have shown that participants with high-risk features by gene array studies tend to have shorter remissions (disappearance of signs and symptoms of myeloma) and do not survive as long as participants with low-risk myeloma. Researchers at MIRT think that one reason for this is that the myeloma cells re-grow in the time when participants are not receiving treatment because they are recovering from high-dose chemotherapy. In this study, participants will receive several chemotherapy drugs previously shown to be effective in myeloma, but in lower doses and in shorter cycles. It is hoped that by giving the drugs in this way, myeloma cells will not have time to re-grow between cycles, therefore resulting in longer remissions. This study is being done in an attempt to improve the remission rate and the survival time for participants with high-risk myeloma.

DETAILED DESCRIPTION:
* To find out if giving multi-agent chemotherapy in lower and more frequent doses to make the timely delivery of chemotherapy cycles possible, will result in better treatment outcomes
* To find out if changing the way the drugs are given during the transplant phase will also result in fewer side effects, while still being effective
* To find out if giving treatment between transplants (called "inter-transplant therapy") will prevent the myeloma from re-growing between transplants
* To find out if long-term maintenance therapy will result in longer remissions
* To find out what the effects (good and bad) of this overall treatment will be
* To learn more about the biology and genetics of multiple myeloma by performing imaging tests and collecting blood, bone marrow aspirate and biopsies, and biopsies of lesions seen on MRI or PET scans for research

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed active MM requiring treatment. Patients with previous history of smoldering myeloma will be eligible if there is evidence of progressive disease requiring chemotherapy.
* Patients must be either untreated o have not had more than one cycle of systemic MM therapy, excluding bisphosphonates and localized radiation.
* Patients must have high-risk disease, as defined by any one of the following:
* GEP risk score of > or = 0.66 or
* LDH > or = 360 U/L Rule out hemolysis, infection an contact PI for clarification
* Zubrod < or = 2, unless solely due to symptoms of MM-related bone disease.
* Patients must have a platelet count of > or = 50,000/uL, unless lower levels are explained by extensive bone marrow plasmacytosis.
* Patients must be at least 18 years of age and not older than 75 years of age at the time of registration.
* Participants must have preserved renal function as defined by a serum creatinine level of < 3 mg/dL.
* Participants must have an ejection fraction by ECHO or MUGA scan > or = 45%
* Patients must have adequate pulmonary function studies > or = 50% of predicted on mechanical aspects (FEV squared, FVC, etc) and diffusion capacity (DLCO) > or = 50% of predicted. If the patient is unable to complete pulmonary function tests due to MM related pain or condition, exception may be granted if the principle investigator documents that the patient is a candidate for high dose therapy.
* Patients must have signed an IRB-approved informed consent indicating their understanding of the proposed treatment and understanding that the protocol has been approved by the IRB.

Exclusion Criteria:

* Does not have high-risk disease
* Poorly controlled hypertension, diabetes mellitus, or other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be acceptable if the patient's life expectancy exceeds five years.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Subjects of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-10; Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Accelerate and sustain, at 2 years from starting therapy | 2 years

SECONDARY OUTCOMES:
48hrs after melphalan 10mg/m2, gene expression profiling (GEP) examinations of CD138-purified MM plasma cells (PC)and of bone marrow biopsy (BX)samples | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, MD, PhD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Ling W, Zangari M, Van Rhee F, Barlogie B, Yaccoby S. Altered mesenchymal and endothelial subsets in interstitial bone marrow and focal lesions in myeloma patients and SCID-hu mice. Haematologica. 2025 Nov 1;110(11):2740-2751. doi: 10.3324/haematol.2025.287717. Epub 2025 Jun 12. PMID 40501401
- [Derived] Pawlyn C. High-risk myeloma: a challenge to define and to determine the optimal treatment. Lancet Haematol. 2021 Jan;8(1):e4-e6. doi: 10.1016/S2352-3026(20)30361-6. Epub 2020 Dec 22. No abstract available. PMID 33357481
- [Derived] Davies FE, Rosenthal A, Rasche L, Petty NM, McDonald JE, Ntambi JA, Steward DM, Panozzo SB, van Rhee F, Zangari M, Schinke CD, Thanendrarajan S, Walker B, Weinhold N, Barlogie B, Hoering A, Morgan GJ. Treatment to suppression of focal lesions on positron emission tomography-computed tomography is a therapeutic goal in newly diagnosed multiple myeloma. Haematologica. 2018 Jun;103(6):1047-1053. doi: 10.3324/haematol.2017.177139. Epub 2018 Mar 22. PMID 29567784
- See also: Multiple Myeloma — http://myeloma.uams.edu/